CLINICAL TRIAL: NCT07177092
Title: Efficacy and Safety of Primary Tumor Resection Combined With Osimertinib in Patients With Advanced EGFR-mutant Non-small Cell Lung Cancer: A Randomized Controlled Study
Brief Title: Primary Tumor Resection Plus Osimertinib in Advanced EGFR-mutant Non-small Cell Lung Cancer
Acronym: SURGAN-TKI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-157-02
Record Dates: First submitted 2025-09-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer; EGFR
Keywords: Non-Small Cell Lung Cancer; EGFR; Randomized controlled trial; Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants will receive oral osimertinib at a dose of 80 mg once daily, continued until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Drug: Osimertinib
- Intervention Group (Experimental): Participants will first undergo cytoreductive surgery. After adequate postoperative recovery for 4-6 weeks, they will receive oral osimertinib at a dose of 80 mg once daily, continued until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Procedure: Surgery; Drug: Osimertinib

INTERVENTIONS:
Procedure: Surgery — ① Preoperative evaluation must confirm resectability. Thoracoscopic minimally invasive surgery will be performed, with the surgical approach selected according to disease conditions, such as lobectomy, segmentectomy, wedge resection, or sleeve resection; ② Systematic mediastinal lymph node dissection or lymph node sampling (based on preoperative imaging and intraoperative evaluation) must be performed; ③ Postoperative recovery must be adequate (postoperative complications ≤ Clavien-Dindo grade II).
  Arms: Intervention Group
Drug: Osimertinib — Dose: 80 mg orally, once daily, until disease progression or the occurrence of unacceptable toxicity. The dose should be administered at approximately the same time each day, at 24-hour intervals.

SUMMARY:
This study is designed to explore whether resecting the primary lung cancer, followed by osimertinib, can improve outcomes for patients with advanced non-small cell lung cancer (NSCLC) harboring sensitizing EGFR mutations (exon 19 deletion or L858R). Patients with stage III-IV NSCLC will be included and randomly assigned to receive either surgery to remove the primary lung cancer followed by osimertinib, or osimertinib alone. All patients will continue treatment until disease progression or they need to stop for another reason. The primary outcome being studied is progression-free survival (PFS). Secondary outcomes include overall survival (OS), objective response rate (ORR), disease control rate (DCR), adverse effects (AEs), serious adverse effects (SAEs) and quality of life (QoL). The findings from this study may help determine whether surgery combined with EGFR tyrosine kinase inhibitor (TKI) provides more benefit than EGFR-TKI alone for patients with EGFR-mutant advanced NSCLC.

DETAILED DESCRIPTION:
Osimertinib is a third-generation EGFR-TKI that has become one of the standard first-line treatments for patients with advanced NSCLC harboring sensitizing EGFR mutations such as exon 19 deletion and L858R substitution. Although osimertinib significantly improves survival outcomes, most patients eventually experience disease progression because of drug resistance, and long-term survival remains limited. Surgical resection has traditionally been reserved for early-stage NSCLC. However, emerging evidence suggests that removing the primary tumor, even in the setting of advanced disease, may help reduce tumor burden, delay resistance, and potentially enhance the effectiveness of systemic therapies. To date, there is little high-quality evidence from randomized trials evaluating the role of primary tumor resection in combination with EGFR-TKI for patients with unresectable stage III-IV NSCLC harboring sensitizing EGFR mutations. This randomized, open-label, phase 2 study is designed to evaluate whether combining primary tumor resection with osimertinib provides superior clinical outcomes compared with osimertinib alone in patients with advanced EGFR-mutant NSCLC. Approximately 118 eligible patients will be randomized in a 1:1 ratio to receive either surgery followed by osimertinib or osimertinib monotherapy. Treatment will continue until disease progression or discontinuation criteria are met. The primary outcome is PFS assessed by independent radiology review according to RECIST v1.1. Secondary outcomes include OS, ORR, DCR, AEs, SAEs and QoL. Statistical analysis will include Kaplan-Meier estimation of median PFS with 95% confidence intervals, log-rank testing for comparing differences between the two treatment groups, and Cox proportional hazards models for calculating hazard ratios. Stratification will be performed based on clinical stage, EGFR mutation type, tumor size, and baseline demographic characteristics. The results of this trial are expected to provide high-level evidence on whether surgery combined with EGFR-TKI offers additional clinical benefit over standard EGFR-TKI alone in advanced EGFR-mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, no restriction on sex.
2. Histologically or cytologically confirmed stage III-IV non-squamous NSCLC, unresectable as assessed by multidisciplinary team (MDT).
3. Presence of EGFR exon 19 deletion (19Del) or L858R mutation, confirmed by ARMS-PCR, NGS, or other validated methods.
4. No prior systemic therapy for lung cancer.
5. ECOG performance status of 0-1.
6. Estimated life expectancy of at least 6 months.
7. Primary lung tumor size ≥1 cm, with at least one measurable lesion remaining after resection according to RECIST v1.1 criteria.
8. Adequate organ function, including:

   ① Hematologic function: absolute neutrophil count ≥1.5 × 10⁹/L; platelet count ≥100 × 10⁹/L; hemoglobin ≥9.0 g/dL.

   ② Hepatic function: ALT and AST ≤2.5 × ULN (≤5 × ULN if liver metastases are present); total bilirubin ≤1.5 × ULN.

   ③ Renal function: serum creatinine ≤1.5 × ULN, or creatinine clearance ≥50 mL/min (Cockcroft-Gault formula).
9. Adequate pulmonary function (must meet at least one of the following to ensure postoperative reserve):

   ① FEV1 ≥1.2 L (or ≥40% of predicted value);

   ② FEV1/FVC ≥0.7, to exclude severe obstructive ventilatory dysfunction;

   ③ DLCO (diffusing capacity for carbon monoxide) ≥40% of predicted value, to assess diffusion capacity.

   ④ If preoperative FEV1 <1.2 L or DLCO <40%, additional cardiopulmonary exercise testing (e.g., 6-minute walk test, stair climbing test) is recommended to evaluate postoperative pulmonary reserve.
10. Evaluated by the study team and deemed suitable for primary tumor resection.
11. Signed written informed consent and willingness to comply with study protocol.

Exclusion Criteria:

1. Presence of any other known EGFR mutations.
2. Histological evidence of mixed small-cell lung cancer (SCLC) or history of transformation to SCLC.
3. Immunodeficiency: history of primary immunodeficiency disorders, or prior allogeneic organ or bone marrow transplantation.
4. Active brain metastases. Patients with adequately treated brain metastases may be eligible if they are neurologically stable for at least 2 weeks before enrollment, and are either not requiring corticosteroids or receiving a stable or decreasing dose of ≤10 mg prednisone (or equivalent) once daily.
5. Pregnancy.
6. Any serious comorbid condition that, in the opinion of the investigator, may interfere with participation in the study or interpretation of study results, including but not limited to: uncontrolled systemic diseases, psychiatric illness, active or uncontrolled infections, or other abnormal findings from laboratory or clinical examinations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | From randomization until the first documentation of disease progression or death from any cause, whichever occurs first (up to 5 years).
  Progression-free survival is defined as the time from randomization to the first documentation of disease progression or death from any cause, whichever occurs first. Disease progression will be assessed by the Independent Radiology Review Committee according to RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival | Randomization to death from any cause (up to 5 years).
  Overall survival is defined as the time from randomization to death from any cause.
Objective Response Rate | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  The proportion of patients achieving complete and partial remission after treatment, measured according to RECIST v1.1 criteria.
Disease Control Rate | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  Disease control rate is defined as the proportion of participants with complete response, partial response, and stable disease, as determined by RECIST v1.1 criteria.
Adverse Events | From randomization to disease progression or death (up to 5 years).
  Safety will be assessed by recording treatment-related adverse events (AEs) and serious adverse events (SAEs), graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of Life (QoL) evaluated by European Organisation for Research and Treatment of Cancer core quality of life questionnaire (EORTC QLQ-C30) | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  The EORTC QLQ-C30 is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients (range: 0-100; higher scores indicate better functioning and quality of life).
Quality of Life (QoL) evaluated by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13) | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  Supplementary lung cancer-specific questionnaire to be used in conjunction with the QLQ-C30 (range: 0-100; higher scores indicate worse lung cancer-related symptoms).

IPD SHARING:
Plan to Share IPD: No